CLINICAL TRIAL: NCT05275803
Title: Clinical and Microbiological Efficacy of Lactobacillus Reuteri as an Adjunctive Therapy to Non-surgical Periodontal Treatment of Chronic Periodontitis With Type 2 Diabetes: a Randomized Controlled Clinical Trial
Brief Title: Lactobacillus Reuteri for Non-surgical Periodontal Treatment of Chronic Periodontitis With Type 2 Diabetes Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Peihui Ding, Associate Professor, The Dental Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DHZhejiangU-2022(025)
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): The participants would use probiotics for 30 days
  Interventions: Dietary Supplement: Probiotics
- Control (Experimental): The participants would use not probiotics
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Probiotics — The participant would receive non-surgical periodontal treatment, after which the participant uses probiotics (BioGaia Prodentis, L. reuteri DSM 17938+L. reuteri ATCC 5289, 0.8g, qn) for another 30 days.
  Arms: Probiotics
Dietary Supplement: Control — The participant does not use probiotics after non-surgical periodontal treatment.
  Arms: Control

SUMMARY:
This study aims to investigate the clinical and microbiological efficacy of Lactobacillus reuteri as an adjunctive therapy to non-surgical periodontal treatment of chronic periodontitis with type 2 diabetes.

DETAILED DESCRIPTION:
Periodontitis and diabetes affect the course and outcome of each other. Many studies have shown that for patients with periodontitis, concomitant diabetes can aggravate the destruction of periodontal tissue and accelerate the progression of periodontitis, which is an important risk factor for periodontitis. Affected by diabetes, patients with poor glycemic control have worse periodontal status, and the prognosis of periodontitis treatment is more suspicious. Conversely, periodontitis also affects diabetic status, and periodontitis is associated with dysglycemia, increased insulin resistance, and increased risk of diabetic complications. After periodontal therapy, it is expected to reduce the level of systemic inflammation and ultimately improve glycemic control and overall prognosis of diabetes. However, the treatment of periodontitis with diabetes is still a challenge, and how to improve the prognosis of patients with periodontitis with type 2 diabetes remains to be studied.

BioGaia Prodentis is a probiotic chewable tablet containing Lactobacillus reuteri (combination of L. reuteri DSM 17938 and L. reuteri ATCC 5289). Studies have shown that the use of the probiotics has an additional effect on periodontal therapy. However, in the periodontitis patients with type 2 diabetes, whether the use of this probiotic can improve the effect of periodontal therapy, few relevant research have published.

ELIGIBILITY:
Inclusion Criteria:

1. age between 35 to 70 years,
2. type 2 diabetes with treatment ≥ 6-month, with HbA1c≤7.5%,
3. generalized periodontitis (Stage III or IV),
4. no less than 15 teeth

Exclusion Criteria:

1. smoking, or quit smoking for less than 5 years;
2. Suffering from other known systemic diseases that can affect the progression of periodontitis (immune abnormalities, osteoporosis, history of head and neck radiotherapy, etc.);
3. Received periodontal treatment within 6 months;
4. Have taken antibiotics, non-steroidal anti-inflammatory drugs, immunosuppressants, hormones and other drugs that affect periodontal within 3 months;
5. Have taken probiotics within 6 months;
6. Prophylactic use of antibiotics is required;
7. Pregnant and lactating women;

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-06-08 (Estimated); Primary Completion 2023-06-20 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
Probing depth | change from baseline to day 90
  measured at six sites of each implant (mesio-labial/buccal, mid-labial/buccal, disto-labial/buccal, mesio-palatal/lingual, mid-palatal/lingual, and disto-palatal/lingual) using a periodontal probe (UNC15)
Microorganism | change from baseline to day 90
  measured by 16s rDNA in subgingival plaque and faces

SECONDARY OUTCOMES:
Gingival index | day 0, 30, 90, 150
  assessed at four sites of each implant (mesio-labial/buccal, mid-labial/buccal, disto-labial/buccal, and palatal/lingual) according to the index of Loe and Silness
Gingival Recession | day 0, 30, 90, 150
  The distance from the implant margin to the gingival margin was measured with a periodontal probe
Bleeding of Probing | day 0, 30, 90, 150
  bleeding after periodontal probing
Fasting Blood Glucose | day 0, 30, 90, 150
  Fasting Blood Glucose in blood
HbA1c | day 0, 30, 90, 150
  HbA1c in blood
IL-1β、IL-6、TNF-α | day 0, 30, 90, 150
  IL-1β、IL-6、TNF-α by ELISA in GCF

IPD SHARING:
Plan to Share IPD: No